CLINICAL TRIAL: NCT02779998
Title: Prophylactic Non-invasive Ventilation During Surgical Procedure in Rhythmology
Acronym: VNI-RYTHMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 38RC15.163
Record Dates: First submitted 2016-05-12; First posted 2016-05-23 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Electrophysiology; Anesthesia; Acute Respiratory Failure
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard oxygen therapy with facial mask (Active Comparator): Patients assigned to standard medical therapy will received supplemental oxygen via a facial Venturi mask at a rate of up to 15 liters per minute in order to maintain peripheral oxygen saturation (SpO2) above 94% during electrophysiology procedure under light sedation.
  Interventions: Other: Standard oxygen therapy with facial mask
- non invasive ventilation (Experimental): non invasive ventilation (NIV) which associated positive end expiratory pressure (PEEP: 5 to 10 cmH2O) and pressure support ventilation (PSV: 5 to 15 cmH2O, to achieve total Pressure bellow 20cmH2O) will be delivered during electrophysiology procedure under light sedation. The patient will received supplemental oxygen through facial mask to achieve an oxygen saturation level above 94%.
  Interventions: Other: non invasive ventilation

INTERVENTIONS:
Other: non invasive ventilation — non invasive ventilation is delivered by a specific respirator with inspiratory help mode. NIV mask and parameters are adapted to obtains a Tidal volume ≤ to 8 ml/kg/cycle (if possible ≤ 6 ml/kg/cycle) and a SpO2 superior of 94%.
  Arms: non invasive ventilation
Other: Standard oxygen therapy with facial mask
  Arms: standard oxygen therapy with facial mask

SUMMARY:
Acute respiratory failure is frequent during rhythmology procedure under light sedation in high risks selected patients. Non invasive ventilation (NIV) is recommended for acute cardiogenic pulmonary oedema and sleep apnea. The investigators will perform a monocentric, prospective, randomized controlled trial to compare the efficacy of NIV which associated pressure support ventilation (PSV: 5 to 15 cmH2O) and positive end expiratory pressure (PEEP: 5 to 10 cmH2O) with standard oxygen therapy in prevention of peroperative respiratory event. Our hypothesis is that peroperative use of NIV should reduce the incidence of apnea and hypoxia during procedure in rhythmology under light sedation.

DETAILED DESCRIPTION:
This study is an investigator-initiated, monocentric, two-arm parallel-group trial with electronic system based randomization. The study protocol was approved by a Central Ethics Committee (France) according to French law. Our teaching hospital have a long experience with peroperative use of NIV during light sedation and acute respiratory failure. This study is designed as a PROBE study (Prospective Randomized Open with Blinded Evaluation) : the investigators will provide a blinded analysis of peroperative computer collected data.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years old or above
* Procedure in electrophysiology laboratory
* High risk patient defined by an American Society of Anesthesiology (ASA) score of 3 or 4

Exclusion Criteria:

* Planned orotracheal intubation
* ASA 1 or 2
* Sleep apnea treated with home non invasive ventilation
* Major contraindication to NIV use
* Pregnancy
* Consent refusal
* Patients protected under the French Law L1121-5 to L1121-8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Respiratory event | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  Based on computer analysis:
  * Hypoxia (pulse oxymetry below 90%)
  * Apnea (No respiratory cycle measured by End-Tidal carbon dioxygen (CO2) for more than 20 seconds)

SECONDARY OUTCOMES:
Occurence of hemodynamic instability | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  Based on computer analysis and defined as: low blood pressure or bradycardia with need of catecholamine drugs or volume resuscitation.
Respiratory rate | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  Based on computer analysis
End-Tidal carbon dioxygen | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  Based on computer analysis
Tidal Volume | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  Based on computer analysis
Respiratory settings of NIV ventilator | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  Based on computer analysis
O2 inspiration fraction | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  Based on computer analysis
Bispectral Index variability | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  Based on computer analysis
Occurence of a major medical event | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  A major medical event is defined as
  * pneumothorax,
  * oro-tracheal intubation or laryngeal mask,
  * cardiopulmonary resuscitation,
  * surgical complication
  * pleural or pericardia effusion drain use
  * Intervention from anesthesiologist
Occurence of a minor medical event | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  A minor medical event is defined as
  * NIV mask related skin injuries,
  * nausea or vomiting,
  * aspiration
  Guedel canula,
  - mandibular subluxation
Procedure failure | during procedure in cardiac electrophysiology laboratory (an average of 2 hours)
  Procedure failure is defined as the change of oxygen device or the change of ventilatory mode (controlled mode)
Patient status | within 7 days after procedure
  A composite outcome defined as the occurence of:
  * death,
  * cardiac complication (acute heart failure, infarcts),
  * acute respiratory failure
  * pneumopathy
Length of hospital stay | within 7 days after procedure
Length of Intensive Care Unit (ICU) stay | within 7 days after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, La Tronche, France

REFERENCES:
- [Derived] Moury PH, Pasquier V, Greco F, Arvieux JL, Alves-Macedo S, Richard M, Casez-Brasseur M, Skaare K, Jacon P, Durand M, Bedague D, Jaber S, Bosson JL, Albaladejo P. A randomized controlled trial of the intraoperative use of noninvasive ventilation versus supplemental oxygen by face mask for procedural sedation in an electrophysiology laboratory. Can J Anaesth. 2023 Jul;70(7):1182-1193. doi: 10.1007/s12630-023-02495-2. Epub 2023 Jun 2. PMID 37268802